CLINICAL TRIAL: NCT05752058
Title: Risk Factors for Early Acute Lung Injury After Liver Transplantation in Children and the Prediction Vaulen
Brief Title: Risk Factors for Early Acute Lung Injury After Liver Transplantation in Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tianjin First Central Hospital (Other)
Responsible Party: Principal Investigator, Yingli Cao, Principal investigator, Tianjin First Central Hospital
Other Study IDs: 2022N105KY
Record Dates: First submitted 2023-02-12; First posted 2023-03-02 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Acute Lung Injury; Liver Transplantation; Risk Factors
Keywords: Acute lung injury; liver transplantation; microRNAs; follistatins-like protein 1; S100A9 protein
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood sample immediately after induction of anesthesia (T1), 10 min at anhepatic stage (T2), 30 min at new hepatic stage (T3) and immediately after abdominal closure (T4)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to identify the risk factors for early acute lung injury (ALI) after liver transplantation in children .The main questions it aims to answer are what the risk factors are for early ALI in children and to evaluate the predictive value for the development of ALI.Participants will be divided into non-ALI group and ALI group according to whether they had ALI in a week after liver transplantation.Researchers will compare the difference between the two groups and use multivariate logistic regression analysis to screen the risk factors of ALI, and receiver operating characteristic(ROC) curve was used to evaluate the predictive efficacy of risk factors.

DETAILED DESCRIPTION:
The goal of this observational study is to identify the risk factors for early acute lung injury (ALI) after liver transplantation in children and evaluate the predictive value for the development of ALI.Perioperative data of patients were obtained through electronic case information management system, anesthesia surgery clinical information system and clinical research database. Basic clinical data of children were recorded, including age, gender, alanine aminotransferase (ALT), aspartate aminotransferase (AST), International Normalized ratio (INR), childhood end-stage liver disease score (PELD) and other indicators.The expression levels of serum microRNA-122, microRNA-21, S100A9,S100A8 ,follistim like protein 1(FSTL1), tumor necrosis factor-α (TNF-α) and interleukin-1β(IL-1β) were recorded immediately after induction of anesthesia (T1), 10 min at anhepatic stage (T2), 30 min at new hepatic stage (T3) and immediately after abdominal closure (T4). Intraoperative fluid intake and outflow, ALT, AST, and serum bilirubin peaks in the first week after surgery were recorded.Murray score was used to determine whether ALI occurred one week after surgery, and the children were divided into non-ALI group and ALI group. Multivariate logistic regression analysis was used to screen the risk factors of ALI, and ROC curve was used to evaluate the predictive efficacy of risk factors.

ELIGIBILITY:
Inclusion Criteria:

* patient was diagnosed with biliary atresia
* American society of anesthesiologists physical status Ⅱ-Ⅲ

Exclusion Criteria:

* Secondary liver transplantation or other important organ injury before surgery
* Present with congenital airway or respiratory malformation
* Acute respiratory infection or respiratory insufficiency was present within 1 month before surgery
* Incomplete data

Ages: 3 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children who needed elective parental liver transplantation due to biliary atresia from January 2020 to December 2022
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
the score of acute lung injury | 1 week after liver transplantation
  Murray score was scored from four aspects: chest X-ray, hypoxemia score, positive end-expiratory pressure and lung compliance. The total score was the sum of the scores of all parameters the sum of the number of parameters adopted. The higher the score, the more serious the injury was.

SECONDARY OUTCOMES:
the expression level of serum microRNA-122,microRNA-21,S100A9,S100A8, TNF-α ,IL-1β and FSTL-1 | immediately after induction of anesthesia (T1), 10 min at anhepatic stage (T2), 30 min at new hepatic stage (T3) and immediately after abdominal closure (T4)
  Real-time fluorescence quantitative polymerase chain reaction (RT-qPCR) was used to detect the expression of microRNA-122,microRNA-21,S100A9,S100A8,TNF-α ,IL-1β and FSTL-1 in serum.

IPD SHARING:
Plan to Share IPD: Undecided